CLINICAL TRIAL: NCT01612377
Title: A Phase II, Double-blind, Controlled, Multi-center, Randomized, Long Term Safety Trial of z102 and Prednisone (5 mg or 7.5 mg) in Patients With Moderate to Severe Rheumatoid Arthritis
Brief Title: Long Term Safety Trial of z102 and Prednisone in Patients With Moderate to Severe Rheumatoid Arthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: missed endpoint of meaningful clinical benefit, compared to prednisolone 2.7mg
Sponsor: Zalicus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Z102-009
Record Dates: First submitted 2012-02-22; First posted 2012-06-05 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Moderate to Severe
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — dipyridamole, prednisolone drug combination; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- prednisolone-dipyridamole (Experimental)
  Interventions: Drug: Prednisolone-Dipyridamole
- prednisone 5mg (Active Comparator)
  Interventions: Drug: Prednisone
- prednisone 7.5mg (Active Comparator)
  Interventions: Drug: prednisone

INTERVENTIONS:
Drug: Prednisolone-Dipyridamole — Oral, QD
  Other Names: Z102
  Arms: prednisolone-dipyridamole
Drug: Prednisone — Oral QD Prednisone 5mg
  Arms: prednisone 5mg
Drug: prednisone — Oral, QD prednisone 7.5mg
  Arms: prednisone 7.5mg

SUMMARY:
This study will compare an experimental drug called Z102 (combination of prednisolone and dipyridamole, against prednisone 5mg and prednisone 7.5mg in patients with moderate to severe Rheumatoid Arthritis for a period of 52 weeks.

DETAILED DESCRIPTION:
This is a long-term Phase II safety study of approximately 52 weeks in duration. Eligible patients will have completed at least 6 weeks of Protocol Z102-008 and will have met all inclusion and exclusion criteria for this study.

All patients will be up-titrated on Z102 over 3 weeks or will receive prednisone 5.0 mg or 7.5 mg:

Primary objectives:

* Adverse events (AEs)
* Vital signs
* Clinical laboratory and clinical chemistry evaluations

Secondary objectives:

* Joint imaging and bone density
* DAS28-CRP and individual components
* Patient Global Assessment of Disease Activity
* American College of Rheumatology criteria (ACR 20, ACR 50, ACR 70)
* Multidimensional Assessment of Fatigue (MAF)
* Time to failure

ELIGIBILITY:
Inclusion Criteria:

* Have completed all 12 weeks of Protocol Z102-008 or discontinued after participating in at least 6 weeks of the randomized withdrawal portion of Z102-008 for acceptable reasons
* Have met all inclusion/exclusion criteria for enrollment into Protocol Z102-008
* Have been on DMARD therapy for at least 90 days and have been on a stable DMARD dose without dosage adjustment or modification for 6 weeks prior to enrollment into Protocol Z102-008, and be able to maintain the same dose of conventional DMARD therapy during Protocol Z102-009 participation

Exclusion Criteria:

* Did not complete 6 weeks of the double-blind section of Protocol Z102-008, or was discontinued from Protocol Z102-008 for reasons of an AE, protocol violation, or non-compliance
* Active cardiovascular disease, unless well controlled by appropriate treatment, for a minimum of 3 months prior to screening for enrollment into Protocol Z102-008
* Currently taking aspirin for reasons other than for cardiovascular prophylaxis or their total daily dose is greater than 325 mg
* Taking oral steroids at a daily prednisone dose, or the equivalent, of >10 mg/day within the past 2 weeks
* Intraarticular, intramuscular, or intravenous glucocorticoids must not have been given at least 6 weeks prior to entering study Protocol Z102-008 or Protocol Z102-009, at any time during the study, or be anticipated to be given at any time during the study
* The need to continue the use of one or multiple NSAIDs at the same time, or use acetaminophen on a chronic basis
* All opiate use is prohibited.
* Use of any other medications or herbs or non-pharmacological treatments (e.g., acupuncture) used for the treatment of pain is prohibited
* Has, or has had, any active severe infections or recent invasive surgical procedures within 30 days of Protocol Z102-008 or Protocol Z102-009 initiation
* HIV, hepatitis B, or hepatitis C infection
* Has undergone administration of any investigational drug within 30 days of study
* All biologic agents are excluded for 90 days prior to Screening and during the conduct of Protocol Z102-008, and Protocol Z102-009
* Has undergone administration of rituximab or any B-cell depleting investigational drugs within 6 months of Protocol Z102-008 Screening or Protocol Z102-009 initiation, or at any time during participation in study Protocol Z102-008
* Has a history of hypersensitivity reaction to glucocorticoids and/or dipyridamole
* Known or suspected history of alcohol or drug abuse within 2 years prior to Screening for Protocol Z102-008
* Has any other medical condition which may interfere with the conduct of this study in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-03; Primary Completion 2013-07 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Difference in incidence rates of adverse events between treament groups | 12 months

SECONDARY OUTCOMES:
Joint imaging | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gene Wright, PHARM.D, PH.D, Study Director — Zalicus, Inc
Locations (1):
- Nemanja Damjanov, Belgrade, Serbia